CLINICAL TRIAL: NCT04215276
Title: Comparison of Valsalva Maneuver and Control in Reducing Pain During Spinal Injection
Brief Title: Valsalva Maneuver and Control in Reducing Pain During Spinal Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Alfan Mahdi Nugroho, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IndonesiaUAnes 048
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Brachytherapy
Keywords: valsalva maneuver; control; pain; spinal injection
MeSH Terms: conditions — Pain | interventions — Valsalva Maneuver

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valsalva Maneuver (Active Comparator): Patient will do valsalva maneuver for 20 seconds
  Interventions: Other: Valsalva maneuver
- control (Placebo Comparator): Patient will do nothing
  Interventions: Other: Control

INTERVENTIONS:
Other: Valsalva maneuver — pressure during Valsalva maneuver was measure using sphygmomanometer
  Arms: Valsalva Maneuver
Other: Control — patient was not given any intervention
  Arms: control

SUMMARY:
The study aimed to compare the effectiveness of Valsalva maneuver as non pharmacological approach and control in reducing pain during spinal injection.

DETAILED DESCRIPTION:
This was an experimental study on 70 subjects with 35 subjects treated with Valsalva maneuver and 35 subjects treated as control from January to April 2019. Research subjects were female who underwent brachytherapy for the first time with spinal anesthesia. The effectiveness in reducing pain was assessed by using Visual Analogue Scale (VAS) and patient movement during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent elective surgery using spinal anesthesia
* patients who have not undergone spinal anesthesia before
* Physical status ASA I or II
* Signing informed consent

Exclusion Criteria:

* have a spinal anesthesia history
* contraindicated for spinal anesthesia
* subjects who cannot do Valsalva to 30mmHg pressure for 20 seconds
* have a allergic history to local anesthetics or opioid drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Pain measurement during injection with VAS score | 30 seconds
  Pain degree was measured with VAS score [0 equals to no pain whereas 10 equals to the maximum pain]

SECONDARY OUTCOMES:
Patient movement | 30 seconds
  Investigator observes patient movement during the first spinal injection

CONTACTS AND LOCATIONS:
Overall Officials: Alfan M Nugroho, MD, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo National Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Calthorpe N. The history of spinal needles: getting to the point. Anaesthesia. 2004 Dec;59(12):1231-41. doi: 10.1111/j.1365-2044.2004.03976.x. PMID 15549987
- [Result] Kumar S, Gautam SK, Gupta D, Agarwal A, Dhirraj S, Khuba S. The effect of Valsalva maneuver in attenuating skin puncture pain during spinal anesthesia: a randomized controlled trial. Korean J Anesthesiol. 2016 Feb;69(1):27-31. doi: 10.4097/kjae.2016.69.1.27. Epub 2016 Jan 28. PMID 26885298
- [Result] Agarwal A, Sinha PK, Tandon M, Dhiraaj S, Singh U. Evaluating the efficacy of the valsalva maneuver on venous cannulation pain: a prospective, randomized study. Anesth Analg. 2005 Oct;101(4):1230-1232. doi: 10.1213/01.ane.0000167270.15047.49. PMID 16192551
- [Result] Cigdem UK, Sevinc S, Esef B, Sureyya O, Muzaffer G, Akif D. [A comparison of three different needles used for spinal anesthesia in terms of squamous epithelial cell transport risk]. Rev Bras Anestesiol. 2017 Sep-Oct;67(5):468-471. doi: 10.1016/j.bjan.2017.04.011. Epub 2017 May 16. Portuguese. PMID 28526468
- [Result] Pstras L, Thomaseth K, Waniewski J, Balzani I, Bellavere F. The Valsalva manoeuvre: physiology and clinical examples. Acta Physiol (Oxf). 2016 Jun;217(2):103-19. doi: 10.1111/apha.12639. Epub 2016 Jan 5. PMID 26662857